CLINICAL TRIAL: NCT03536754
Title: A Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Study to Evaluate the Safety and Efficacy of CCX140-B in Subjects With Focal Segmental Glomerulosclerosis (FSGS)
Brief Title: A Study of CCX140-B in Subjects With FSGS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CL011_140; LUMINA-1 (Other: Chemocentryx); NCT03536754 (Other: US NCT number); 134007 (Other: IND)
Record Dates: First submitted 2018-03-28; First posted 2018-05-25 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: FSGS; Focal Segmental Glomerulosclerosis; Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — CCX140-B

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, Phase 2
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Placebo Comparator): Placebo (N=10)
  Interventions: Other: Placebo
- Group B (Experimental): CCX140-B 5 mg once daily (N=10)
  Interventions: Drug: CCX140-B
- Group C (Experimental): CCX140-B 10 mg twice daily (N=10)
  Interventions: Drug: CCX140-B
- Group D (Experimental): CCX140-B 15 mg twice daily (N=10)
  Interventions: Drug: CCX140-B

INTERVENTIONS:
Other: Placebo — Three placebo tablets, taken twice daily (BID), per os, for 84 days (12 weeks)
  Other Names: CCX140-B Placebo
  Arms: Group A
Drug: CCX140-B — One 5 mg CCX140-B tablet and 2 placebo tablets in the morning; 3 placebo tablets in the evening; per os, for 84 days.
  Other Names: Group B
  Arms: Group B
Drug: CCX140-B — Two 5 mg CCX140-B tablets and 1 placebo tablet, taken BID; per os, for 84 days.
  Other Names: Group C
  Arms: Group C
Drug: CCX140-B — Three 5 mg CCX140-B tablets, taken BID; per os, for 84 days.
  Other Names: Group D
  Arms: Group D

SUMMARY:
A Multicenter, Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Study to Evaluate the Safety and Efficacy of CCX140-B in Subjects with FSGS to be conducted in the North America, Europe and Australia

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Study to Evaluate the Safety and Efficacy of CCX140-B in Subjects with Focal Segmental Glomerulosclerosis (FSGS) to be conducted in the North America, Europe and Australia. The aim of this study is to evaluate the effect of treatment with CCX140-B, a selective antagonist of C-C chemokine receptor type 2 in subjects with focal segmental glomerulosclerosis on urinary protein excretion as assessed by changes in urine protein to creatinine ratio (UPCR).

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-75
2. UPCR ≥ 1 g protein/g creatinine (or at 113 mg.mmol) at screening
3. Diagnosis of FSGS based on renal biopsy or high risk genetic variant
4. Diagnosis of one of primary FSGS based on characteristic histopathology, medical history and clinical course or FSGS secondary to genetic variants associated with increased risk or severity.
5. Estimated glomerular filtration rate (eGFR) >30 mL/min/1.73m2
6. Clinical stable blood pressure not to exceed 145/95 mmHg
7. RAAS blockers must be stable for at least 4 weeks prior to screening and projected to remain stable through week 12, unless adjustments are required for management of hypertension.
8. Immunosuppressive or immunomodulatory therapy must be stable for at least 4 weeks prior to screening and projected to remain stable through study week 12
9. Glucocorticoids must be stable for at least 4 weeks prior to screening and projected to remain stable through study week 12.
10. Both genders of childbearing potential must agree to use adequate contraception during and for at least 3 months after the last dose of study drug.
11. Subjects must be willing and able to give written Informed Consent and to comply with protocol requirements.
12. Subjects must be judged to be otherwise fit for the study by the Investigator. -

Exclusion Criteria:

1. Pregnant or nursing
2. History of organ transplantation
3. On an organ transplant waiting list or anticipated organ transplant within 6 months of screening
4. Anti-CD20 monoclonal antibodies within 20 months of screening are exclusionary. Subjects that used anti CD20 monoclonal antibodies prior to week 20 are allowed with confirmed recovery of CD20+ B cell population to within normal range
5. Plasmapheresis within 12 weeks of screening
6. BMI ≥40
7. Participation in any clinical study of an investigational product within 12 weeks or 5 half-lives of screening
8. Currently on dialysis or likely to require dialysis during the blinded treatment phase of the study.
9. History or presence of any form of cancer within 5 years of screening except excised basal cell or squamous cell carcinoma or carcinoma in situ such as cervical or breast carcinoma in situ that has been excised or completed resected without evidence or recurrence.
10. Positive HBV, HCV, or HIV viral screening test. Subjects who have received highly effective therapy for HCV demonstrated to have negative viral titers for at least 6 months following discontinuation of treatment, will be considered to have a negative HCV screening test
11. Renal disease associated with disorders other than FSGS that is active or has significant risk of progressing during the course of the study.
12. Disorders that are associated with FSGS lesions.
13. Evidence of tuberculosis.
14. Evidence of hepatic disease with the exception that isolated INR elevation in the absence of other significant liver enzyme abnormalities is explained by anticoagulant therapy, (e.g. warfarin)
15. Hematologic abnormalities as follows: Hb <8 g/dL, platelets <50,000, ANC <1000 cells/µL) at baseline.
16. QTcF greater than 450 msec.
17. History of alcohol or illicit drug abuse or of lithium, pamidronate and interferon. Recreational use of cannabis is not excluded where legal.
18. History of gastrointestinal conditions that may interfere with study medication compliance.
19. Known hypersensitivity to CCX140-B or inactive ingredients of the CCX140-B tablets (including microcrystalline cellulose, starch, crospovidone, magnesium stearate, or silicon dioxide).
20. History or presence of systemic disorder other than FSGS that requires, or is expected to require, systemic glucocorticoids or immune modulators during the study; topical or inhaled glucocorticoids and immune modulators are not excluded.
21. History or presence of any medical condition or disease which, in the opinion of the Investigator, may place the subject at unacceptable risk for study participation.
22. Subjects taking strong CYP3A4 inducers or strong CYP3A4 inhibitors within two weeks prior to screening.
23. Subjects taking lithium or interferon; subjects taking non-steroidal anti-inflammatory agents (NSAIDS) chronically (intermittent, i.e. occasional NSAIDS for pain or fever is discouraged, but is not excluded).

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (37):
- United States (9):
  - AKDHC, Phoenix, Arizona
  - Los Angeles Biomedical Research Institute, Torrance, California
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - MGH, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - East Carolina University, Greenville, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Health Sciences Center, Houston, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
- Australia (3):
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville
- Canada (4):
  - St. Josephs Healthcare - Hamilton, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre (Odette Cancer Center), Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CISSS de la Monteregie-Centre - Hopital Charles LeMoyne, Greenfield Park, Quebec
- France (5):
  - CHU Bordeaux- Hospital Pellegrin, Bordeaux
  - CHU Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - APHM - Hopital de la Conception, Marseille
  - Hopitaux Prives de Metz, Metz
- Italy (5):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - IRCCS Azienda Ospedaliera Universitaria San Martino IST, Genova
  - Presidio Ospedaliero di Montichiari-A.O. Spedali Civili di Brescia, Montichiari
  - Fondazione S. Maugeri IRCCS, Pavia
  - Fondazione Policlinico Universitario A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
- New Zealand (2):
  - North Shore Hospital, Takapuna, Auckland
  - Taranaki Base Hospital, New Plymouth
- Poland (5):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku - II Klinika Nefrologii z Oddzialem Leczenia Nadcisnienia Tetniczego i Pododdzialem Dializoterapii, Bialystok
  - SCM Sp. Zo.o., Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnez Centralny Szpital, Lodz
  - Samodzielny Publiczny Szpital Kliniczny, Szczecin
  - Uniwersytecki Szpital Kliniczny Klinika Nefrologii i Medycyny Transplantacyjnej, Wroclaw
- United Kingdom (4):
  - Cambridge University - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Salford Royal NHS Foundation Trust Manchester, Salford
  - Morriston Hospital, Swansea

REFERENCES:
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment took place in Australia, Canada, France, Italy, New Zealand, Poland, United Kingdom, and in the United States. The target was to enroll 40 male or female subjects. The first patient was enrolled on 17 May 2018. A total of 84 subjects were screened; 38 subjects failed screening and 46 subjects were randomized.
Pre-assignment Details: Eighty-four (84) patients were screened. Screen failure occurred in 38 (45.2%) subjects due to not meeting inclusion or exclusion criteria (35 [41.7%] subjects) and other reasons (3 [3.6%] subjects).
Groups:
- Placebo: Placebo: Placebo
- CCX140-B 5 mg Once Daily: CCX140-B 5 mg once daily
  CCX140-B: CCX140-B is an orally administered selective antagonist of CCR2
- CCX140-B 10 mg Twice Daily: CCX140-B 10 mg twice daily
  CCX140-B: CCX140-B is an orally administered selective antagonist of CCR2
- CCX140-B 15 mg Twice Daily: CCX140-B 15 mg twice daily
  CCX140-B: CCX140-B is an orally administered selective antagonist of CCR2
- Open-label Extension: Following the 12-week Blinded Treatment Period, all subjects who remained eligible took open-label CCX140-B for an additional 12 weeks (84 consecutive days) at the highest tolerated dose under evaluation, which was determined to be 15 mg BID.
Period: Double Blind Period 1
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Started | 12 | 11 | 12 | 11 | 0
Completed | 12 | 11 | 11 | 11 | 0
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Period: Open Label Extension
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Started | 0 (46 subjects were randomised in Period A. Only 43 subjects entered the Open-Label Extension.) | 0 (46 subjects were randomised in Period A. Only 43 subjects entered the Open-Label Extension.) | 0 (46 subjects were randomised in Period A. Only 43 subjects entered the Open-Label Extension.) | 0 (46 subjects were randomised in Period A. Only 43 subjects entered the Open-Label Extension.) | 43
Completed | 0 | 0 | 0 | 0 | 42
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo control
- Total: Total of all reporting groups
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Total
Number analyzed (Participants) | 12 | 11 | 12 | 11 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 11 | 10 | 44
  >=65 years | 0 | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Screening
  years | 46.3 (12.50) | 41.7 (12.70) | 37.9 (15.51) | 43.4 (13.26) | 42.3 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 3 | 16
  Male | 8 | 7 | 7 | 8 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 11 | 10 | 11 | 9 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 11 | 10 | 11 | 9 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
UPCR at screening [Count of Participants; unit: Participants] — UPCR (Urine protein g:creatinine g) Urine protein:creatinine ratio (g protein/g creatinine) ≥3.5 Units (g/dL)
  Participants
    UPCR ≥ 3.5 at screening | 3 | 2 | 3 | 3 | 11
    UPCR < 3.5 at screening | 9 | 9 | 9 | 8 | 35
UPCR at baseline [Number; unit: g/dL] — UPCR (Urine protein g:creatinine g)
  g/dL
    UPCR ≥ 3.5 at baseline | 1 | 1 | 3 | 4 | 9
    UPCR < 3.5 at baseline | 11 | 10 | 9 | 7 | 37
Concomitant use of ACE inhibitor or ARB or aldosterone antagonists [Count of Participants; unit: Participants] — ACE - Angiotensin-converting enzyme ARB - Angiotensin receptor blockers
  Participants
    Yes | 12 | 10 | 11 | 10 | 43
    No | 0 | 1 | 1 | 1 | 3
Current use of glucocorticoids and/or immunosuppressive medications [Count of Participants; unit: Participants]
  Yes | 7 | 6 | 6 | 6 | 25
  No | 5 | 5 | 6 | 5 | 21
Concomitant use of glucocorticoids [Count of Participants; unit: Participants]
  Yes | 6 | 4 | 4 | 5 | 19
  No | 6 | 7 | 8 | 6 | 27
Concomitant use of all calcineurin inhibitors combined [Count of Participants; unit: Participants] — Includes cyclosporin or tacrolimus
  Participants
    Yes | 2 | 4 | 3 | 3 | 12
    No | 10 | 7 | 9 | 8 | 34
Concomitant use of calcineurin inhibitors cyclosporin [Count of Participants; unit: Participants]
  Yes | 1 | 1 | 3 | 1 | 6
  No | 11 | 10 | 9 | 10 | 40
UPCR [Mean (Standard Deviation); unit: g protein/g creatinine] — UPCR - urine protein:creatinine ratio
  g protein/g creatinine | 2.19 (1.029) | 2.00 (1.149) | 2.86 (2.008) | 3.12 (2.504) | 2.54 (1.773)
Baseline eGFR (CKD-EPI Creatinine-Cystatin C) [Mean (Standard Deviation); unit: ml/min/1.73 m^2] — Baseline estimated Glomerular Filtration Rate (Chronic Kidney Disease Epidemiology Collaboration Creatinine-Cystatin C)
  ml/min/1.73 m^2 | 72.75 (36.204) | 56.18 (28.927) | 54.67 (15.622) | 61.36 (32.265) | 61.35 (29.163)
Baseline urine MCP-1 creatinine ratio [Mean (Standard Deviation); unit: g protein/g creatinine] — Baseline urine MCP-1 creatinine ratio MCP-1: monocyte chemoattractant protein 1
  g protein/g creatinine | 453.74 (438.384) | 576.41 (470.089) | 504.02 (388.569) | 430.66 (325.651) | 490.67 (399.559)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in UPCR at Week 12
Description: Least squared mean ratio of UPCR (Urine protein g:creatinine g) compared to baseline at Week 12 in the ITT population. ITT- Intent to treat
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (90% Confidence Interval); unit: g protein/g creatinine
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 11 | 11
g protein/g creatinine | 0.83 [0.69 to 0.99] | 1.02 [0.84 to 1.23] | 1.12 [0.93 to 1.35] | 0.87 [0.72 to 1.05]
Statistical Analysis 1: Comparison: Placebo vs CCX140-B 5 mg Once Daily; Test type: Superiority; p = 0.1924, Mixed effects model for repeated measure — ≤ 0.1924; LSM Ratio = 1.23, 90% CI 2-sided [0.95 to 1.6], Standard Error of Mean 1.171
Statistical Analysis 2: Comparison: Placebo vs CCX140-B 10 mg Twice Daily; Test type: Superiority; p = 0.0612, Mixed effects model for repeated measure — ≤ 0.0612; LSM Ratio = 1.35, 90% CI 2-sided [1.04 to 1.76], Standard Error of Mean 1.172
Statistical Analysis 3: Comparison: Placebo vs CCX140-B 15 mg Twice Daily; Test type: Superiority; p = 0.7653, Mixed effects model for repeated measure — ≤ 0.7653; LSM Ratio = 1.05, 90% CI 2-sided [0.81 to 1.36], Standard Error of Mean 1.169
Statistical Analysis 4: Comparison: Placebo vs CCX140-B 5 mg Once Daily vs CCX140-B 10 mg Twice Daily vs CCX140-B 15 mg Twice Daily; Test type: Superiority; p = 0.1537, Mixed effects model for repeated measure — ≤ 0.1537; LSM Ratio = 1.2, 90% CI 2-sided [0.97 to 1.48], Standard Error of Mean 1.136

2. Primary Outcome: Number of Participants of Treatment-emergent AEs (TEAE), TEAEs Leading to Study Withdrawal, and Serious Adverse Events (SAEs)
Description: TEAEs leading to study withdrawal means study drug discontinuation in this endpoint.
Time Frame: Baseline to Week 12, and Week 12 to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 12 | 11 | 43
Participants
  TEAEs | 10 | 6 | 8 | 7 | 24
  SAEs | 0 | 0 | 0 | 0 | 1
  TEAEs leading to study withdrawal | 0 | 0 | 1 | 0 | 2

3. Primary Outcome: Change From Baseline in Activated Partial Thromboplastin Time
Description: Normal Range: 23.9 - 40.0
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Population: Data is not available for all participants.
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 10 | 10 | 10 | 40
second
  Week 12 | 2.40 (4.259) | 2.05 (4.396) | 2.36 (2.614) | 1.28 (2.508) | 1.76 (4.332)
  Week 24: number analyzed (Participants) | 11 | 10 | 10 | 9 | 40
  Week 24 | 2.91 (4.132) | 1.39 (3.187) | 2.34 (6.169) | 0.10 (3.223) | 1.76 (4.332)

4. Primary Outcome: Change From Baseline in Plasma Alanine Aminotransferase
Description: Normal Range: 6 - 41 U/L
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
U/L | 0.5 (2.70) | 0.8 (5.22) | 0.3 (3.29) | -1.8 (2.95) | 0.0 (3.65)

5. Primary Outcome: Change From Baseline in Plasma Alkaline Phosphatase
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
U/L | 10.2 (7.08) | -1.0 (11.59) | 0.7 (15.86) | -1.9 (9.45) | 2.3 (12.16)

6. Primary Outcome: Change From Baseline in Plasma Amylase
Description: Normal range: 22-123 U/L
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
U/L | 3.1 (16.11) | 8.9 (18.30) | 5.0 (24.56) | 3.9 (23.19) | 5.2 (20.09)

7. Primary Outcome: Change From Baseline in Plasma Aspartate Aminotransferase
Description: Normal range : 9-34 U/L
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
U/L | 18.3 (6.17) | -0.4 (4.60) | -3.5 (7.71) | -3.2 (3.07) | -1.7 (5.25)

8. Primary Outcome: Change From Baseline in Plasma Bicarbonate
Description: Normal range: 21-33 mmol/L
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mmol/L | 0.5 (3.45) | -0.4 (3.24) | 0.9 (3.59) | -0.6 (2.83) | 0.1 (3.24)

9. Primary Outcome: Change From Baseline in Plasma Bilirubin
Description: Normal range: 0.1-1.10 mg/dL
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 0.044 (0.1985) | -0.006 (0.2796) | 0.160 (0.2381) | -0.012 (0.1519) | 0.050 (0.2263)

10. Primary Outcome: Change From Baseline in Plasma C Reactive Protein
Description: Normal range: 0.0-3.0 mg/L
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/L | 1.200 (3.1597) | 2.144 (8.5528) | -1.000 (4.6448) | -1.444 (3.8014) | 0.260 (5.4276)

11. Primary Outcome: Change From Baseline in Plasma Calcium
Description: Normal range: 8.5-10.5 mg/dL
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 0.18 (0.387) | 0.20 (0.427) | 0.17 (0.498) | -0.01 (0.454) | 0.14 (0.434)

12. Primary Outcome: Change From Baseline in Plasma Chloride
Description: Normal range: 95-110 mmol/L
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mmol/L | -0.5 (2.70) | 0.9 (1.79) | -0.8 (3.31) | 3.2 (2.33) | 0.6 (2.97)

13. Primary Outcome: Change From Baseline in Plasma Cholesterol
Description: Normal range: 100-200 mg/dL
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | -2.7 (31.11) | -2.0 (27.67) | 18.9 (48.17) | -43.0 (64.17) | -5.6 (47.99)

14. Primary Outcome: Change From Baseline in Plasma Creatine Kinase
Description: Normal range: 23-210 U/L
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
U/L | 21.2 (39.65) | 18.1 (59.20) | -19.5 (89.93) | 14.2 (206.95) | 11.9 (89.15)

15. Primary Outcome: Change From Baseline in Plasma Creatinine
Description: Normal range: 0.62-1.44 mg/dL
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 41
mg/dL | 0.060 (0.1437) | 0.033 (0.2461) | 0.115 (0.2186) | 0.147 (0.3790) | 0.161 (0.3926)

16. Primary Outcome: Change From Baseline in Plasma Cystatin C
Description: Normal range: 0.53-0.95 mg/L
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/L | 0.114 (0.1838) | 0.104 (0.1074) | 0.093 (0.2896) | 0.018 (0.2198) | 0.087 (0.2436)

17. Primary Outcome: Change From Baseline in Plasma Direct Bilirubin
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 0.011 (0.0396) | 0.008 (0.0316) | 0.005 (0.0497) | -0.005 (0.0254) | 0.004 (0.0373)

18. Primary Outcome: Change From Baseline in Plasma Glucose
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 40
mg/dL | -5.3 (15.11) | 1.1 (10.58) | 1.5 (16.91) | -6.2 (14.07) | -0.9 (14.27)

19. Primary Outcome: Change From Baseline in Plasma HDL Cholesterol
Description: HDL -High-density lipoprotein
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 0.8 (5.75) | -2.3 (12.95) | 2.1 (20.41) | 2.4 (9.65) | 0.7 (9.39)

20. Primary Outcome: Change From Baseline in Plasma Indirect Bilirubin
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 0.043 (0.1033) | -0.009 (0.0919) | 0.054 (0.2866) | -0.043 (0.1572) | 0.046 (0.1947)

21. Primary Outcome: Change From Baseline in Plasma LDL Cholesterol
Description: LDL - Low-density lipoprotein
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 10 | 11 | 10 | 10 | 38
mg/dL | 12.2 (19.97) | -2.8 (11.36) | 8.0 (24.86) | -8.9 (37.78) | -5.0 (37.61)

22. Primary Outcome: Change From Baseline in Lactate Dehydrogenase
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
U/L | -10.2 (25.67) | -26.4 (69.73) | -14.5 (26.09) | 5.1 (27.15) | -12.0 (41.83)

23. Primary Outcome: Change From Baseline in Plasma Pancreatic Lipase
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
U/L | 3.6 (9.71) | 8.1 (24.14) | -5.2 (9.81) | 24.5 (51.50) | 9.0 (50.27)

24. Primary Outcome: Change From Baseline in Plasma Magnesium
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 0.10 (0.148) | 0.02 (0.140) | -0.02 (0.240) | 0.09 (0.321) | 0.01 (0.199)

25. Primary Outcome: Change From Baseline in Plasma Phosphate
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 0.33 (0.609) | 0.16 (0.423) | 0.15 (0.596) | 0.04 (0.803) | 0.04 (0.580)

26. Primary Outcome: Change From Baseline in Plasma Potassium
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 38
mmol/L | 0.09 (0.327) | 0.12 (0.232) | -0.09 (0.305) | 0.23 (0.789) | 0.00 (0.514)

27. Primary Outcome: Change From Baseline in Plasma Protein
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
g/dL | 0.17 (0.320) | 0.05 (0.305) | -0.11 (0.575) | -0.09 (0.396) | 0.00 (0.515)

28. Primary Outcome: Change From Baseline in Prothrombin Intl. Normalised Ratio
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: Prothombin intl. normalised ratio
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 10 | 10 | 10 | 40
Prothombin intl. normalised ratio | 0.03 (0.210) | 0.01 (0.160) | 0.10 (0.141) | 0.01 (0.088) | 0.08 (0.387)

29. Primary Outcome: Change From Baseline in Prothrombin Time
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 10 | 10 | 10 | 40
second | 0.48 (1.566) | 0.07 (1.561) | 0.69 (1.268) | 0.33 (0.736) | 0.78 (3.445)

30. Primary Outcome: Change From Baseline in Plasma Sodium
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mmol/L | 0.0 (2.22) | 1.8 (3.89) | 0.9 (3.59) | 2.5 (5.05) | 1.0 (3.46)

31. Primary Outcome: Change From Baseline in Plasma Triglycerides
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 16.6 (123.84) | 5.7 (51.48) | -16.5 (25.80) | -23.2 (123.79) | -2.6 (80.08)

32. Primary Outcome: Change From Baseline in Plasma Urate
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 0.51 (0.485) | 0.04 (1.107) | -0.28 (0.877) | -0.08 (0.926) | -0.05 (1.040)

33. Primary Outcome: Change From Baseline in Plasma Urea Nitrogen
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 41
mg/dL | 2.8 (3.65) | -2.6 (4.18) | 3.6 (5.95) | 1.1 (11.42) | 2.3 (6.15)

34. Primary Outcome: Change From Baseline in Basophils
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
cells x 10^9/L | 0.02 (0.058) | 0.03 (0.047) | 0.02 (0.60) | -0.03 (0.048) | 0.02 (0.063)

35. Primary Outcome: Change From Baseline in Basophils/Leukocytes
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: percentage of basophils in leukocytes
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
percentage of basophils in leukocytes | 0.08 (0.389) | -0.01 (0.459) | 0.18 (0.547) | -0.13 (0.419) | 0.16 (0.433)

36. Primary Outcome: Change From Baseline in Eosinophils
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 12 | 11 | 39
cells x 10^9/L | 0.01 (0.108) | 0.01 (0.122) | 0.00 (0.184) | 0.01 (0.099) | 0.03 (0.162)

37. Primary Outcome: Change From Baseline in Eosinophils/Leukocytes
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: percentage of Eosinophils in Leukocytes
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
percentage of Eosinophils in Leukocytes | 0.32 (1.375) | 0.09 (0.984) | -0.02 (2.245) | 0.33 (1.430) | 0.27 (1.922)

38. Primary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular HGB Concentration
Description: HGB - Hemoglobin
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
g/dL | -0.20 (0.603) | -0.18 (0.778) | -0.24 (0.439) | -0.16 (0.556) | -0.28 (0.891)

39. Primary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Hemoglobin
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: picogram(s)
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
picogram(s) | -0.2 (0.58) | -0.3 (0.47) | -0.5 (0.82) | 0.0 (0.82) | -0.1 (0.80)

40. Primary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
fL | -0.21 (1.472) | -0.02 (2.093) | -0.33 (1.251) | 0.03 (1.931) | 0.44 (1.801)

41. Primary Outcome: Change From Baseline in Erythrocytes
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: cells x 10^12/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
cells x 10^12/L | -0.004 (0.2946) | 0.055 (0.2211) | 0.010 (0.2326) | -0.55 (0.1761) | -0.003 (0.2968)

42. Primary Outcome: Change From Baseline in Hematocrit
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in blood
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
percentage of red blood cells in blood | -0.3 (2.34) | 0.5 (2.11) | -0.1 (2.26) | -0.8 (1.55) | 0.2 (2.61)

43. Primary Outcome: Change From Baseline in Hemoglobin
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
g/dL | -0.12 (0.802) | 0.13 (0.588) | -0.10 (0.784) | -0.25 (0.488) | -0.07 (0.923)

44. Primary Outcome: Change From Baseline in Leukocytes
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: cells x 10^3/microlitre
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
cells x 10^3/microlitre | -0.98 (1.915) | 0.45 (1.012) | 0.37 (1.819) | -0.09 (1.928) | -0.09 (1.711)

45. Primary Outcome: Change From Baseline in Lymphocytes
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: cells x 10^3/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
cells x 10^3/L | -0.080 (0.2152) | 0.122 (0.3541) | 0.099 (0.4865) | 0.194 (0.9257) | 0.161 (0.4165)

46. Primary Outcome: Change From Baseline in Lymphocytes/Leukocytes
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes in leukocytes
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
percentage of lymphocytes in leukocytes | 2.51 (5.052) | 0.06 (6.287) | -0.99 (8.132) | 1.52 (7.013) | 2.61 (7.099)

47. Primary Outcome: Change From Baseline in Monocytes/Leukocytes
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: percentage of monocytes in leukocytes
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
percentage of monocytes in leukocytes | 1.38 (1.641) | 0.25 (2.056) | 0.99 (3.022) | 0.56 (1.532) | -0.21 (2.262)

48. Primary Outcome: Change From Baseline in Neutrophils
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: cells x 10^3/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
cells x 10^3/L | -0.954 (1.6290) | 0.255 (1.1041) | 0.137 (1.6023) | -0.289 (1.4171) | -0.281 (1.5104)

49. Primary Outcome: Change From Baseline in Neutrophils/Leukocytes
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: percentage of neutrophils in leukocytes
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
percentage of neutrophils in leukocytes | -4.28 (5.941) | -0.39 (6.548) | -0.16 (8.247) | -2.28 (7.230) | -2.84 (7.830)

50. Primary Outcome: Change From Baseline in Platelets
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 10 | 11 | 10 | 43
cells x 10^9/L | 5.2 (31.68) | 26.2 (30.10) | 4.8 (28.72) | 0.9 (27.65) | 19.1 (54.30)

51. Primary Outcome: Change From Baseline in Reticulocytes/Erythrocytes
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: percentage of reticulocytes/erythrocytes
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 39
percentage of reticulocytes/erythrocytes | -0.08 (0.626) | -0.11 (0.554) | -0.30 (0.615) | -0.12 (0.290) | -0.14 (0.536)

52. Primary Outcome: Change From Baseline in Urine Albumin
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 42
mg/dL | 1.117 (118.7664) | -19.044 (119.7149) | -8.455 (53.9332) | -35.964 (178.9164) | -28.433 (107.8847)

53. Primary Outcome: Change From Baseline in Urine Creatinine
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 42
mg/dL | 10.65 (35.931) | -11.67 (33.432) | -15.37 (30.920) | 25.30 (84.654) | -6.96 (31.530)

54. Primary Outcome: Change From Baseline in Urine Protein
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 42
mg/dL | -19.3 (139.96) | -8.9 (134.17) | -9.0 (80.51) | -80.6 (230.57) | -35.1 (144.93)

55. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 12 and Week 24
Description: Change from baseline in eGFR calculated by the CKD-EPI Cystatin C equation, CKD-EPI Creatinine equation, CKD-EPI Creatinine-Cystatin C equation and MDRD Creatinine equation at Weeks 12 and 24. CKD-EPI: Chronic Kidney Disease Epidemiology Collaboration; MDRD: Modification of Diet in Renal Disease Open label extension covers Baseline to Week 12 and Baseline to Week 24
Time Frame: Baseline to Week 12 (double-blind treatment period) and Week 12 to Week 24 (open-label extension)
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 43
mL/min/1.73 m^2
  CKD-EPI Cystatin C equation Week 12 | -4.9 (11.74) | -3.1 (3.91) | -1.6 (8.61) | 0.2 (9.51) | -1.7 (9.49)
  CKD-EPI Cystatin C equation Week 24 | -0.8 (6.63) | -3.2 (10.40) | -1.3 (9.69) | -3.2 (9.60) | -2.0 (8.86)
  CKD-EPI Creatinine equation Week 12 | -3.0 (6.47) | -4.2 (11.50) | -3.9 (5.74) | -4.8 (9.68) | -4.7 (9.68)
  CKD-EPI Creatinine equation Week 24 | -3.1 (5.74) | -8.2 (9.89) | -5.3 (10.59) | -2.0 (8.29) | -4.7 (8.80)
  CKD-EPI Creatinine-Cystatin C equation Week 12 | -5.3 (8.92) | -3.5 (5.61) | -2.6 (6.53) | -2.8 (8.57) | -3.2 (8.43)
  CKD-EPI Creatinine-Cystatin C equation Week 24 | -2.4 (5.24) | -5.5 (9.20) | -3.2 (9.18) | -2.8 (7.93) | -3.4 (7.82)
  MDRD Creatinine equation Week 12 | -4.7 (10.82) | -5.1 (13.75) | -4.6 (6.23) | -6.7 (14.03) | -5.6 (13.76)
  MDRD Creatinine equation Week 24 | -4.5 (11.12) | -8.8 (12.85) | -5.9 (10.05) | -4.0 (10.77) | -5.8 (10.95)

56. Secondary Outcome: Proportion of Subjects Achieving Complete or Partial Renal Remission at Week 12 and Week 24
Description: 1. Proportion of subjects achieving complete renal remission by the following definition at Weeks 12 and 24 o Reduction in UPCR to <0.3 g/g o Serum albumin within normal range (for subjects with abnormal serum creatinine levels at baseline, return to normal levels for that age group; for subjects with normal serum creatinine levels at baseline, final value within 20% of baseline levels) 2. Proportion of subjects achieving partial remission defined as UPCR reduction of ≥50% from baseline and UPCR <3.5 g/g (definition 1), assessed at Weeks 12 and 24 3. Proportion of subjects achieving partial remission defined Decrease in UPCR to less than 1.5 g/g and at least a 40% reduction in proteinuria from baseline (definition 2), assessed at Weeks 12 and 24
Time Frame: Endpoint at Week 12 for Double-Blind Treatment Period and Endpoint at Week 24 for Open-Label Extension
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CCX140-B 5 mg Once Daily | CCX140-B 10 mg Twice Daily | CCX140-B 15 mg Twice Daily | Open-label Extension
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 43
Participants
  Complete renal remission | 0 | 0 | 0 | 0 | 0
  Partial remission (definition 1) | 1 | 0 | 0 | 1 | 4
  Partial remission (definition 2) | 0 | 0 | 0 | 0 | 6

ADVERSE EVENTS:
Time Frame: From Baseline to Week 24
Groups:
- CCX140-B 5 mg: CCX140-B 5 mg once daily
  CCX140-B: CCX140-B is an orally administered selective antagonist of CCR2
- CCX140-B 10 mg: CCX140-B 10 mg once daily
  CCX140-B: CCX140-B is an orally administered selective antagonist of CCR2
- CCX140-B 15 mg: CCX140-B 15 mg once daily
  CCX140-B: CCX140-B is an orally administered selective antagonist of CCR2
- Placebo Open Label: Placebo control
  For Period B of trial
- CCX140-B 5mg Open Label: CCX140-B 5 mg once daily
  CCX140-B: CCX140-B is an orally administered selective antagonist of CCR2 For Period B of trial
- CCX140-B 10mg Open Label: CCX140-B 10 mg once daily
  CCX140-B: CCX140-B is an orally administered selective antagonist of CCR2 For Period B of trial
- CCX140-B 15mg Open Label: CCX140-B 15 mg once daily
  CCX140-B: CCX140-B is an orally administered selective antagonist of CCR2 For Period B of trial
Arm/Group | Placebo | CCX140-B 5 mg | CCX140-B 10 mg | CCX140-B 15 mg | Placebo Open Label | CCX140-B 5mg Open Label | CCX140-B 10mg Open Label | CCX140-B 15mg Open Label
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/11 | 0/11 | 0/11 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/11 | 0/11 | 0/11 | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 7/11 | 8/11 | 10/12 | 8/11 | 7/11 | 6/11 | 6/11 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | CCX140-B 5 mg (N=11) | CCX140-B 10 mg (N=12) | CCX140-B 15 mg (N=11) | Placebo Open Label (N=11) | CCX140-B 5mg Open Label (N=11) | CCX140-B 10mg Open Label (N=11) | CCX140-B 15mg Open Label (N=10)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | CCX140-B 5 mg (N=11) | CCX140-B 10 mg (N=12) | CCX140-B 15 mg (N=11) | Placebo Open Label (N=11) | CCX140-B 5mg Open Label (N=11) | CCX140-B 10mg Open Label (N=11) | CCX140-B 15mg Open Label (N=10)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 4 (5) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 2 (3) | 2 (4) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (5) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (2) | 1 (6) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grip strength decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immunosuppressant drug level increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystatin C increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03536754/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT03536754/SAP_001.pdf